CLINICAL TRIAL: NCT02165696
Title: Effectiveness of the Combination of Compression Bandaging and Manual Lymph Drainage in Women With Secondary Lymphedema After Breast Cancer.
Brief Title: Compression Bandaging and Manual Lymph Drainage in Women With Lymphedema
Acronym: LYMPHATIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, Ph D, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMA_CBM_2014/LYMP; Lymphatic Multimodal Treatment
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Arm Lymphedema After Breast Cancer
Keywords: compression bandage, manual lymphatic drainage, lymphedema, breast cancer, qualitative research.
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Manual Lymphatic Drainage; Combined Modality Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual lymphatic drainage and compression bandaging (Experimental): Experimental group: 30 minutes and one hour maximum time of manual lymphatic drainage and compression bandaging with multilayer inelastic bandages with low extensibility. It is possible to apply bandages two or three times per week. Also, an elastic bandage is also held in hand fingers with slight compression and other protective bandage is used in skin. The treatment will be carried out for six weeks five days a week
  Interventions: Other: Multimodal treatment: compression bandaging and manual lymph drainage.
- Manual lymphatic drainage (Active Comparator): Control group: 30 minutes and one hour maximum time of manual lymphatic drainage. The treatment will be carried out for six weeks five days a week.
  Interventions: Other: Manual lymph drainage

INTERVENTIONS:
Other: Multimodal treatment: compression bandaging and manual lymph drainage. — 30 minutes and one hour maximum time of manual lymphatic drainage and compression bandaging with multilayer inelastic bandages with low extensibility. It is possible to apply bandages two or three times per week. Also, an elastic bandage is also held in hand fingers with slight compression and other protective bandage is used in skin. The treatment will be carried out for six weeks five days a week
  Other Names: Multimodal treatment
  Arms: Manual lymphatic drainage and compression bandaging
Other: Manual lymph drainage — 30 minutes and one hour maximum time of manual lymphatic drainage. The treatment will be carried out for six weeks five days a week.
  Arms: Manual lymphatic drainage

SUMMARY:
Lymphedema is the result of accumulation of fluid and other elements in tissue spaces because of an imbalance between the production of fluid interstitial and transport. Lymphedema can cause significant physical and psychological morbidity. Prevalence of lymphedema in patients after breast cancer surgery is 12-60% and the incidence is 12-26%.Psychological and social consequences of secondary lymphedema related breast cancer have been little recognized and documented. Although, it have performed many studies related secondary lymphedema it not found sufficient evidence in the literature to suggest the most effective treatment. There is some evidence suggesting that compression therapy and manual lymphatic drainage can improve lymphedema but more studies are needed. The aim of this research is to to evaluate the clinical effect of multimodal treatment (compression bandaging and manual lymph drainage) versus applying manual lymphatic drainage in women with arm lymphedema after breast cancer surgery.

DETAILED DESCRIPTION:
This study has two sub research: a quantitative approach and a qualitative approach. The research will be carried out by a multicenter way

Quantitative approach consist in carried out a single-blind randomized controlled trial of 44 women with arm lymphedema. Patients will be distributed in two intervention groups by a randomized way. Participants will be given his assignment by closed envelope. Both treatments will be administered five days a week for six weeks. The experimental group (n=22) will receive multimodal treatment: combination of manual lymphatic drainage and compression bandaging. The control group (n=22) only will receive manual lymphatic drainage. We want to determinate the effect on volume arm decrease, quality of life, level of hand strength, degree of pain, fatigue level, and state of anxiety and depression. The influence on the lymphedema will be analyzed with lower limbs strength, physical activity, lung function, respiratory muscle strength by maximal inspiratory and expiratory pressure measurements (MIP and MEP) and cardiorespiratory functional capacity. Patients adherence will be analyzed by a smartphone.

Qualitative apprach: to know the perceptions and experiences of the participants in both interventions groups through a qualitative descriptive study. Data will be obtained with semi-structured depth interview.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 65 years with secondary lymphedema in upper limb after breast cancer surgery.
* Cancer stages I-III according to TNM classification of the American Joint Committee on Cancer.

Exclusion Criteria:

* To have received lymphedema treatment previously.
* To be treated by radiation therapy or chemotherapy.
* Distant metastases or local recurrence of cancer.
* Infectious signs in the upper limb with lymphedema.
* Uncontrolled hypertension.
* Heart disease.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Perimetry | Baseline, 6 weeks and 12 weeks
  Arm volume is measured with perimetry through truncation of cones formula

SECONDARY OUTCOMES:
Handgrip strength | Baseline, 6 weeks and 12 weeks
  Handgrip strength will be determined using hydraulic hand dynamometer "JAMAR"
Multiple sit-to-stant test | Baseline, 6 weeks and 12 weeks
  Multiple sit-to-stant test will be used to evaluate lower limbs strength.
Degree of pain | Baseline, 6 weeks and 12 weeks
  The degree of pain in the affected side with lymphedema will be measured by digital algometer "Commander ™"
Pulmonary function test | Baseline, 6 weeks and 12 weeks
  Simple spirometry to measure lung function with a spirometer "DATOSPIR120"
Maximal inspiratory pressures (MIP) and maximal expiratory pressures (MEP) | Baseline, 6 weeks and 12 weeks
  The strength of the respiratory muscles is measured through a digital manovacuometer (DATOSPIR120)
Six-minute walking test | Baseline, 6 weeks and 12 weeks
  Cardiorespiratory functional capacity as measured with six-minute walking test.
FACT-B+4 questionnaire | Baseline, 6 weeks and 12 weeks
  FACT-B+4 questionnaire to measure quality of life in patients with breast cancer and lymphedema. Alpha of cronbach: 0,52-0,92
EORTIC-QLQ-C30 questionnaire | Baseline, 6 weeks and 12 weeks
  EORTIC-QLQ-C30 questionnaire measures the quality of life in cancer. Alpha of cronbach: 0,52 y 0,89
QLQ BR23 questionnaire | Baseline, 6 weeks and 12 weeks
  QLQ BR23 questionnaire to know quality of life in patients with breast cancer. Alpha of cronbach: 0,48 y 0,94
HADS questionnaire | Baseline, 6 weeks and 12 weeks
  HADS questionnaire to measure depression and anxiety. Alpha of cronbach: 0´8-0´76
QuickPIPPER questionnaire | Baseline, 6 weeks and 12 weeks
  QuickPIPPER questionnaire measures the level of fatigue in breast cancer. Alpha of cronbach: 0,730- 0,961
The short version of the IPAQ | Baseline, 6 weeks and 12 weeks
  The short version of the IPAQ questionnaire for physical activity level. Alpha of cronbach: 0,75
Qualitative measures | 6 weeks
  Data collection was carried out through an interview in-depth semi-structured. The dimensions of the study were developed based on bibliography and objectives of the study: perceptions and experiences with multimodal treatment, ways of living with lymphedema, life style, Physical activity and exercise.
Smartphone-based application | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks
  Smartphone-based application to analyze the treatment adherence of the participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Málaga, Málaga, Málaga, Spain